CLINICAL TRIAL: NCT00805506
Title: Evaluation of Glucose Monitoring Methods: Characterizing Glycemic Control in Subjects With Diabetes
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); LifeScan (Industry)
Responsible Party: Roger S. Mazze, PhD, International Diabetes Center
Other Study IDs: 03349-05-A
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes
Keywords: continuous glucose monitoring accuracy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes Insulin Treated: People with type 1 or type 2 diabetes on insulin.

SUMMARY:
Evaluate the usefulness of continuous glucose monitoring devices in terms of their ability to identify periods throughout the day when glucose varies significantly.

DETAILED DESCRIPTION:
Many CGM systems use a surrogate for blood glucose--tissue glucose or interstitial glucose. Interstitial fluid (ISF) is the medium for these approaches. A physiological lag in ISF glucose relative to capillary blood glucose has been noted, probably due to relatively low blood perfusion at the sampling site. 9 This physiological lag can result in an accuracy error, manifesting as a significant bias between blood and tissue glucose, particularly during periods of rapid glucose change. This lag error might be particularly meaningful when glucose is rapidly dropping towards hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* adult
* A1c >7.4 within last 4 months
* type 1 or 2 diabetes treated with basal/bolus insulin

Exclusion Criteria:

* under 18 years of age
* unable to read/write english
* allergy to adhesives
* employee of CGM company

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with diabetes who are treated with insulin
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To collect sufficient glucose data by means of continuous glucose monitoring for the purpose of detecting clinically relevant alterations in blood glucose throughout a typical or modal day. | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Mazze, PhD, Principal Investigator — International Diabetes Center at Park Nicollet; Elinor (Ellie) S Strock, APRN BC, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States